CLINICAL TRIAL: NCT00742495
Title: A Phase I/II Pharmacokinetic Study of Intravenous and Oral Forodesine in Children With Relapsed or Refractory T-cell or B-cell Precursor Acute Lymphoblastic Leukaemia or T-cell Non-Hodgkin's Lymphoma.
Brief Title: Pharmacokinetic Study of Forodesine in Children With Relapsed or Refractory T-cell or B-cell Precursor Acute Lymphoblastic Leukaemia or T-cell Non- Hodgkin's Lymphoma.
Acronym: BCX1777-108
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow Recruitment
Sponsor: Mundipharma Research Limited (Industry)
Collaborators: Innovative Therapies For Children with Cancer Consortium (Other)
Responsible Party: Mundipharma Research Ltd, Mundipharma Research Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCX1777-108; 2008-00221942
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-02

CONDITIONS: Relapsed or Refractory T-cell Acute Lymphoblastic Leukaemia; B-cell Precursor Acute Lymphoblastic Leukaemia; T-cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Recurrence; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell | interventions — forodesine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Forodesine — PK study

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, pharmacodynamics and safety of different doses of intravenous and oral Forodesine in children with relapsed or refractory T-cell or B-cell precursor Acute Lymphoblastic Leukaemia or T-cell Non-Hodgkin's Lymphoma. Preliminary efficacy will also be assessed.

DETAILED DESCRIPTION:
A multi-centre, multi-national, open label trial of Forodesine in children with relapsed or refractory T-cell or B-cell precursor Acute Lymphoblastic Leukaemia or T-cell Non-Hodgkin's Lymphoma. The primary objective of the study is to evaluate the pharmacokinetics and pharmacodynamics of six different dose schedules of Forodesine. Secondary objectives are to evaluate safety and to collect preliminary efficacy data. All patients will receive active drug. The Initial Treatment Phase will last 37 days with a final response assessment on Day 37. Patients who achieve a response may be eligible to receive extended treatment with Forodesine for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥ 2 years to ≤18 years. ≥ 13 kg
* Female subjects of childbearing potential (i.e. have reached the age of menarche) must have a negative serum or urine pregnancy test recorded prior to the first dose of study medication, be non-lactating, and be willing to use adequate and highly effective method of contraception throughout the study and for one month after the last dose of study medication, if sexually active.
* Sexually active male subjects must be willing and able to use a barrier form of contraception (i.e. condoms) or sexual abstinence throughout the study and for one month after the last dose of study medication
* Unequivocal histological diagnosis of T-ALL, BCP-ALL or T-NHL (World Health Organisation [WHO] classification) at initial diagnosis
* Relapse (³25% marrow blasts) or failure to respond after at least one standard regimen for their disease for subjects with a T-cell malignancy who are ineligible for other therapy of greater curative potential, or failure to respond after at least two standard regimens for subjects with a B-cell precursor malignancy
* KPS or LPS (as appropriate for subject's age) scores ³60
* Anticipated life expectancy of at least 6 weeks
* Adequate kidney (creatinine levels ≤ 2.0 times upper limit of normal) and liver function tests (aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT] ≤3 times upper limit of normal and total bilirubin ≤5 times upper limit of normal)
* Signed ICF and assent if appropriate according to local laws and regulations prior to start of any study specific procedures.

Exclusion criteria:

* Females who are pregnant (positive β-hCG test) or lactating
* Subjects with a history of HIV and/or HTLV-1
* Subjects with known active HBV, HCV, CMV and/or EBV infection
* Subjects with clinical evidence of active symptomatic CNS disease
* Subjects with active serious infection
* Prior treatment with any antileukemic agent, chemotherapy or leukophoresis treatment within 7 days (within 4-5 days for 6-mercaptopurine (MP) and within 2 days for low-dose methotrexate) prior to study entry
* Lack of full recovery from adverse drug reactions due to prior therapy, independent of when that therapy was given
* Concurrent treatment with other anticancer agents (CNS prophylaxis e.g. intrathecal methotrexate and corticosteroid use will not be excluded)
* Subjects who have chronic gastrointestinal disease or conditions that may hamper compliance and/or absorption of the product; however, study drug administration via nasogastric or gastrostomy tube is allowed
* Any history of hypersensitivity or intolerance to any component of the study medication.
* Subjects who have received an investigational medicinal product within 30 days of study entry (defined as the start of the Screening Period).
* Current participation in another clinical trial is not permitted unless the sole purpose of the trial is for long term follow up/survival data.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2009-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics and pharmacodynamics - data will be collected on Day 1, 5, 8 and 36. | Day 1, and 36

SECONDARY OUTCOMES:
Safety data will be collected throughout the study. Efficacy will be assessed on Day 15 and Day 37. | Day 15 and 37

CONTACTS AND LOCATIONS:
Locations (6):
- Vienna, Austria
- Prague, Czechia
- Prof Gerard Michel, Marseille, France
- Charite Universitymedicine, Berlin, Germany
- Dr Giovanna Gioriani, Pavia, Italy
- Sally Kinsey, Leeds, United Kingdom